CLINICAL TRIAL: NCT04483232
Title: Achromobacter Spp: Description of Epidemiology and Resistance in Chronic Ear Infections and in Healthy Individuals.
Acronym: AERIO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: AMOUREUX FPA 2020
Record Dates: First submitted 2020-07-17; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Achromobacter; Epidemiology; Chronic Ear Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects
  Interventions: Biological: Ear canal swab
- Patients with ear infections
  Interventions: Biological: Ear canal swab

INTERVENTIONS:
Biological: Ear canal swab — Ear canal swab

SUMMARY:
Hearing loss can be the result of chronic ear infections. The role of bacteria of the genus Achromobacter is not known in these conditions. An epidemiological study including a large number of patients is needed to compare the prevalence of these bacteria in sick and healthy subjects, and to highlight the characteristics of the strains and the factors favouring their emergence.

ELIGIBILITY:
Inclusion Criteria:

* Person or parent who has given his or her non-opposition
* Person over 10 years of age
* Sick Subjects Group :

diagnosis of chronic infection by an ENT specialist doctor if patient already included: new episode > 3 months after the complete clinical recovery from the previous episode observed by the ENT doctor - Healthy group: no ear infection in the last 6 months and no antibiotics in the previous month.

Exclusion Criteria:

-

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Protected adult (curatorship, guardianship)
  * Person deprived of their liberty by judicial or administrative decision
  * Pregnant, parturient or breastfeeding woman
  * Adult unable to give consent
  * For healthy subjects:
    * current ear infection or within the last 6 months
    * Antibiotics (local or systemic) taken within the previous month
  * For sick subjects who have already been included once, new episode < 3 months after the previous one
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Achromobacter positive sample number | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France